CLINICAL TRIAL: NCT03218631
Title: Pharmacokinetics of a Medium Chain Triglyceride Oil Oxandrolone Solution vs. Tablets in Healthy Adults: A Relative Bioavailability Study
Brief Title: Oxandrolone in Healthy Adults: A Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Phillip Burch, MD, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99086
Record Dates: First submitted 2017-04-04; First posted 2017-07-14 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Bioavailability
Keywords: oxandrolone, cardiac
MeSH Terms: interventions — Oxandrolone

STUDY DESIGN:
Intervention Model Description: 1. Male
  2. Age 18 to 35 years (inclusive) at the time of screening
  3. Body mass index [BMI, body weight (kg)/height (m)2] below 30 kg/m2
  4. Medically healthy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxandrin (Other): Administration of a single dose of approximately 0.1 mg/kg of a medium chain triglyceride (MCT) oil Oxandrin (oxandrolone) solution vs. 01.mg/kg tablets in a small cohort of healthy adults. Participants will be dosed at two time points one week apart.
  Interventions: Drug: Oxandrin

INTERVENTIONS:
Drug: Oxandrin — The primary outcome for this study will be measurements of the pharmacokinetics of a single dose of oxandrolone 0.1 mg/kg both in tablet form and in the MCT oil preparation. Blood samples for pharmacokinetics will be drawn at 9 timepoints.
  Safety will be assessed by recording adverse events and assessment of hepatic function at baseline and one week following oxandrolone dosing.
  Other Names: Oxandrolone

SUMMARY:
To assess the pharmacokinetics and relative bioavailability of a single dose of approximately 0.1 mg/kg of a medium chain triglyceride (MCT) oil oxandrolone solution vs. tablets in a small cohort of healthy adults.

DETAILED DESCRIPTION:
The results of this study will provide data regarding the relative bioavailability of a novel preparation of oxandrolone in MCT oil, which will allow dosing in neonates and small infants. This pilot study will provide information to design a larger multicenter study of neonates undergoing surgery for complex congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age 18 to 35 years (inclusive) at the time of screening
3. Body mass index [BMI, body weight (kg)/height (m)2] below 30 kg/m2
4. Medically healthy

Exclusion Criteria:

1. Known allergy to anabolic steroids
2. Use of any prescription medication currently or within 14 days prior to dosing
3. Use of tobacco or nicotine containing products (including smoking cessation products), within 6 months prior to dosing
4. Any chronic medical condition
5. Seated blood pressure <90/40 mmHg or >140/90 mmHg at screening
6. Heart rate <40 or >99 at screening
7. Subjects who have taken any investigational drug within 30 days prior to first dose in the current study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects will be included to avoid the possibility of a pregnant female inadvertently receiving the study drug and to eliminate any cofounders related to gender. Oxandrolone is contraindicated in pregnancy. Subjects will be enrolled without regard to race and ethnicity.
Enrollment: 6 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) curve | Measurement of Peak Plasma Concentration (Cmax) at 15 min, 30 min, 1, 2, 3, 4, 8, 24, 48 hours on Days 1 and 8
  The primary outcome for this study will be the pharmacokinetics of a single dose of oxandrolone 0.1 mg/kg both in tablet form and in the MCT oil preparation as measured by peak plasma concentration (Cmax) curve
Area under the plasma concentration versus time curve (AUC) | Measurements at 15 min, 30 min, 1, 2, 3, 4, 8, 24, 48 hours on Days 1 and 8
  The primary outcome for this study will be the pharmacokinetics of a single dose of oxandrolone 0.1 mg/kg both in tablet form and in the MCT oil preparation as measured by the area under the plasma concentration versus time curve (AUC).

SECONDARY OUTCOMES:
Safety will be assessed by recording adverse events and assessment of hepatic function at baseline and one week following oxandrolone dosing. | Liver function will be assessed by measuring serum transaminase levels at baseline and 1 week after each oxandrolone dose in the study participants, and any adverse events throughout the study period and up to 1 week after final dosing will be recorded.
  The risks associated with the 2 doses of oxandrolone given during the course of this study are minimal. Known adverse effects of anabolic steroids, including hepatic dysfunction and virilization, are typically associated with longer-term use (months of daily dosing) and are very unlikely to occur in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip T. Burch, MD, Principal Investigator — University of Utah
Locations (1):
- Primary Children's Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Individual Patient data will only be shared with the research team